CLINICAL TRIAL: NCT02884388
Title: Effects of a Combined Nerve Block on Intraoperative Stress and Postoperative Immune Function in Elderly Patients Subjected to Total Hip Replacement: Study Protocol for a Randomized Controlled Trial
Brief Title: A Combined Nerve Block in Elderly Patients Subjected to Total Hip Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qinghai University (Other)
Responsible Party: Principal Investigator, Liangde A, Associate Chief Physician, Qinghai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QinghaiUH_002
Record Dates: First submitted 2016-08-19; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Arthropathy of Hip
MeSH Terms: interventions — Anesthesia, General; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental group (Experimental): Combined nerve block will be used, involving lower lumbar plexus, sciatic nerve, and paraspinal nerve L1-2.
  Interventions: Procedure: combined nerve block
- control group (Experimental): General anesthesia will be used in this group.
  Interventions: Procedure: general anesthesia

INTERVENTIONS:
Procedure: combined nerve block — Patients in this group were assigned to receive lower lumbar plexus block, sciatic nerve block, and paraspinal nerve L1-2 block.
  Other Names: experimental group
  Arms: experimental group
Procedure: general anesthesia — Patients in this group were assigned to receive general anesthesia.
  Other Names: control group
  Arms: control group

SUMMARY:
The purpose of this study is to validate the hypothesis that a combined nerve block produces better outcomes including intraoperative stress, hemorrheological indexes, postoperative immune function, and incidence of postoperative complications than general anesthesia.

DETAILED DESCRIPTION:
The elderly patients have poor tolerance to anesthesia and total hip replacement because of severe surgical trauma and much blood loss. General anesthesia is a primary anesthesia method used previously for total hip replacement in the elderly and it has many limitations, for example, it can interfere with the physiological function in the elderly patients. The organic function and compensative ability of the elderly are often weakened to varying degrees because of cardiovascular disease, pulmonary disease or diabetes mellitus, thus nociceptive stimuli such as anesthesia and surgery greatly influence the stress.

Stress refers to an organism's non-specific reactions to various nociceptive stimuli, i.e., stressors, in which many factors are involved. It can stimulate sympathetic nerves, strengthen the function of hypothalamic-pituitary-adrenal axis, and cause changes in various metabolisms, thereby playing an important role in maintaining intraoperative vital signs and recovering postoperative immune function. Different anesthesia methods produce different effects on organism's immune function. Effects of anesthesia on immune function are closely related to the complications, such as postoperative infection. In addition, the immunity in the elderly is relatively poorer than that in the normal healthy population. Therefore, a rational anesthesia method is of important clinical significance for safe surgery and postoperative recovery in the elderly. A combined nerve block has been reportedly to be more suitable for total hip replacement in the elderly because of its safety and reliability.

Previous related studies focused primarily on onset time of anesthesia and postoperative complications. To the best of our knowledge, no studies have been reported on the effect of a combined nerve block on intraoperative stress and postoperative immune function in the elderly patients subjected to total hip replacement. Therefore, this study is innovative in our mind.

Adverse events

If severe adverse events including any expected or unexpected symptoms occur, information including the data of occurrence, type of adverse events, measures taken related to the treatment of the adverse events will be reported to the project manager and the institutional review board within 24 hours.

Data collection, management, analysis and open access

Data collection: according to trial design type and requirement, a table will be developed to record trial data. The recorded data will be input into an electronic database using a double-data entry strategy by trained professional staff.

Data management: information accuracy will be checked when all recruited patients are followed up. The database will be locked by the researcher in charge and will not be altered. All information relating to this trial will be preserved by Qinghai University Affiliated Hospital, China.

Data analysis: The electronic database will be made available to a professional statistician for statistical analysis. An outcome analysis report will be made by the statistician and submitted to the lead researchers. An independent data monitoring committee will supervise and manage the trial data with the goal of ensuring a scientific and stringent trial process, resulting in accurate and complete data.

Data open access: Anonymized trial data will be published at http://www.figshare.com.

Statistical analysis

Statistical analysis will be performed by a statistician using SPSS 19.0 software and will follow the intention-to-treat principle. Normally distributed measurement data will be expressed as a mean, standard deviation, min, and max. Non-normally distributed measurement data will be expressed as a lower quartile (q1), median, and upper quartile (q3).

The Mann-Whitney U test will be used to compare fasting blood glucose level, serum cortisol concentration, hemorrheological indexes and immune function-related indices between experimental and control groups. The Mcnemar χ2 test will be used to compare the incidence of adverse events between experimental and control groups, with an accepted significance level of α = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Blood pressure below 160/90 mmHg (1 mm = 0.133 kPa)
* Hemoglobin > 90 g/L
* Fasting blood glucose level < 10 mM
* Preoperative examinations (blood, urine, stool tests, hepatic and renal function, blood coagulation, electrolyte level and electrocardiogram): normal
* Type I-II in American Society of Anesthesiology (ASA) classification
* Age > 65 years
* Of either sex
* Provision of signed informed consent to participate in the trial

Exclusion Criteria:

* Severe heart, liver, lung, kidney or hematological system diseases, severe infection or malignant tumor
* Allergy to anesthetic agents
* Are taking immunosuppressive agents and/or glucocorticoid
* Viral infections
* Mental disorder, dysnoesia, hearing disorder or poor compliance during the anesthesia
* Alcohol or drug abuse

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Intraoperative serum cortisol concentration | during surgery
  To evaluate intraoperative stress response. The normal serum cortisol concentration is 138-635 nM measured at 8:00 a.m.-10:00 a.m. and 83-359 nM at 4:00 p.m.-6:00 p.m. Greater intraoperative serum cortisol concentration indicates stronger stress response.

SECONDARY OUTCOMES:
Serum cortisol concentration | prior to anesthesia, prior to and immediately after surgery
  to evaluate patient's stress response.
Blood glucose level | prior to anesthesia, prior to, during and immediately after surgery
  to evaluate patient's stress response at each time period. The fasting blood glucose in the normal population is 3.61-6.11 mM. Higher fasting blood glucose level indicates stronger stress response .
Incidence of adverse events | 1, 3, 7 days and 3 months after surgery
  These adverse events include upper respiratory tract infection, pulmonary infection, acute atelectasis and acute pulmonary embolism.

CONTACTS AND LOCATIONS:
Overall Officials: Liangde A, Master, Principal Investigator — Affiliated Hospital of Qinghai University
Locations (1):
- Qinghai University Affiliated Hospital, Xining, Qinghai, China

IPD SHARING:
Plan to Share IPD: Undecided